CLINICAL TRIAL: NCT03648619
Title: Evaluation of an Innovative Automatized "Semi-Whole-Body"-MRI Protocol to Increase Patient Comfort and Cost-effectiveness of Oncologic Imaging
Brief Title: Automatized "Semi-Whole-Body"-MRI Protocol for Cancer Staging
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient recruitment
Sponsor: Kantonsspital Baden (Other)
Responsible Party: Principal Investigator, Daniel Hausmann, Head of Abdominal and Oncologic Imaging, Kantonsspital Baden
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2017-00964
Record Dates: First submitted 2018-08-23; First posted 2018-08-27 (Actual); Last update posted 2021-09-09 (Actual); Status verified 2021-09

CONDITIONS: Oncology
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: Clinically-indicated PET/CT and additional study-related MRI as a single Intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Oncologic patients (Other): Oncologic patients with a previous PET/CT for whole-body staging
  Interventions: Diagnostic Test: Semi whole-body MRI

INTERVENTIONS:
Diagnostic Test: Semi whole-body MRI — Single semi-automatic, semi whole-body MRI protocol (Dot engine)

SUMMARY:
The aims of this study are

* to evaluate the image quality and robustness of a whole-body MRI protocol by using an innovative partially automatic algorithm (DOT engine), that automatically optimizes protocol parameters depending on body region (e.g. thorax versus abdomen)
* to compare lesion detectability between wb-MRI and the gold standard positron emission tomography (PET)/CT
* to compare patient comfort between PET/CT and wb-MRI using a dedicated questionnaire
* to compare duration of image acquisition with regards to cost-effectiveness

DETAILED DESCRIPTION:
Whole-body imaging becomes increasingly important in oncologic patients not only for primary cancer staging, but also for assessment of response to therapy. So far, PET/CT is a key method to assess cancer-related changes of metabolism in tumors, which is crucial for response evaluation and to differentiate between benign and malignant lesions. Limitations of PET/CT include the assessment of sclerotic bone metastasis, which often do not show increased tracer uptake. Certain organ metastasis (especially in brain and liver) are also barely detectable due to physiologically increased uptake. Moreover, both CT and administration of radioactive tracer are associated with radiation exposure for patients. Whole-body MRI (wb-MRI) including functional techniques (e.g. Diffusion-weighted Imaging (DWI) to evaluate cell density) enables a functional staging and therapy assessment without use of ionizing radiation. Advantages to assess sclerotic bone lesions and organ metastases have been confirmed in recent literature. Limitations of MRI include detection of lesions in organs with high susceptibility and motion like the thorax.

ELIGIBILITY:
Inclusion Criteria:

* Clinically indicated PET/CT for cancer staging or response assess-ment in patients with histopathologically confirmed solid tumors (e.g.prostate, breast, gastrointestinal, testicles)
* MRI can be scheduled within 1 week to PET/CT exam

Exclusion Criteria:

* general MRI contraindications (devices (e.g. certain pacemakers), pregnancy, claustrophobia)
* severely reduced general condition
* impaired renal function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2018-09-01 (Actual)

PRIMARY OUTCOMES:
to compare lesion detectability between wb-MRI and the gold standard PET/CT | 30 minutes duration of study-related MRI protocol
  - Primary outcome will be the organ based malignant lesion detectability (Thorax, Abdomen). This will be quantified as a dichotomous variable (present/absent) for MRI and PET/CT.
  Outcome will be based on two board certified radiologists. In case of disagreement, consensus will be taken. Results will be obtained in a single reading after inclusion of 50 patients. Readers will be blinded to clinical patient data and results of PET/CT.

SECONDARY OUTCOMES:
Secondary outcome will be the number of lesions | 5 minutes assessment of a dedicated questionnaire to assess patient comfort
  Secondary outcome will be the number of lesions (Hereby, more than 5 lesions per organ will be regarded as diffuse organ involvement (e.g. diffuse bone metastasis)). Moreover, subjective image perception (e.g. image quality (1-5), quality of lesion demarcation (1-3), diagnostic confidence (1-3) will be assessed. A dedicated questionnaire to assess patient comfort and compare patient acceptance of MRI and PET/CT will be evaluated.

CONTACTS AND LOCATIONS:
Locations (1):
- Kantonsspital Baden, Institute of Radiology, Baden, Canton of Aargau, Switzerland

IPD SHARING:
Plan to Share IPD: No